CLINICAL TRIAL: NCT05363397
Title: Safety and Tolerability of Adjunctive TBO-309 in Reperfusion for Stroke
Acronym: STARS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Florey Institute of Neuroscience and Mental Health (Other)
Collaborators: Neuroscience Trials Australia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: CCD78277; U1111-1270-5195 (Other: World Health Organization (WHO) Universal Trial Number (UTN))
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke
Keywords: Antiplatelet therapy; Stroke; Blood clot; Intravenous thrombolysis (IVT); Endovascular Thrombectomy (EVT); TBO-309
MeSH Terms: conditions — Ischemic Stroke; Stroke; Thrombosis

STUDY DESIGN:
Intervention Model Description: Continual Reassessment Method
Who Masked: Outcomes Assessor
Masking Description: Independent imaging assessors will review and adjudicate blinded study data to ensure the primary endpoint meets consistent pre-determined diagnostic criteria. This will include centralised review of de-identified CT and MRI/MRA images. Members will be qualified physicians who are independent of the study and not involved in study management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TBO-309 30mg (25% of target dose) (Experimental): Following randomisation, 30mg TBO-309 will be administered at the same time as the rt-PA infusion or tenecteplase bolus (as part of intravenous thrombolysis) or as soon as practical.
  The allocated dose of TBO-309 will be given intravenously as follows:
  * 20% of the dose will be administered as a bolus over approximately one minute; then
  * the remainder of the dose (80%) will be administered over 3 hours as an infusion
  Only one dose will be administered to the patient.
  Interventions: Drug: TBO-309
- TBO-309 60mg (50% of target dose) (Experimental): Following randomisation, 60mg TBO-309 will be administered at the same time as the rt-PA infusion or tenecteplase bolus (as part of intravenous thrombolysis) or as soon as practical.
  The allocated dose of TBO-309 will be given intravenously as follows:
  * 20% of the dose will be administered as a bolus over approximately one minute; then
  * the remainder of the dose (80%) will be administered over 3 hours as an infusion
  Only one dose will be administered to the patient.
  Interventions: Drug: TBO-309
- TBO-309 120mg (100% of target dose) (Experimental): Following randomisation, 120mg TBO-309 will be administered at the same time as the rt-PA infusion or tenecteplase bolus (as part of intravenous thrombolysis) or as soon as practical.
  The allocated dose of TBO-309 will be given intravenously as follows:
  * 20% of the dose will be administered as a bolus over approximately one minute; then
  * the remainder of the dose (80%) will be administered over 3 hours as an infusion
  Only one dose will be administered to the patient.
  Interventions: Drug: TBO-309
- TBO-309 180mg (150% of target dose) (Experimental): Following randomisation, 180mg TBO-309 will be administered at the same time as the rt-PA infusion or tenecteplase bolus (as part of intravenous thrombolysis) or as soon as practical.
  The allocated dose of TBO-309 will be given intravenously as follows:
  * 20% of the dose will be administered as a bolus over approximately one minute; then
  * the remainder of the dose (80%) will be administered over 3 hours as an infusion
  Only one dose will be administered to the patient.
  Interventions: Drug: TBO-309

INTERVENTIONS:
Drug: TBO-309 — TBO-309 is a potent, selective and ATP competitive PI3Kβ inhibitor which blocks platelet activation adhesion/aggregation and promotes platelet disaggregation, thereby specifically inhibiting thrombosis without interfering with normal haemostasis.

SUMMARY:
STARS is a prospective, multicentre, open-label, dose escalation, Phase IIa study to assess the safety and tolerability of TBO-309, an adjuvant antiplatelet therapy, in patients with AIS.

Acute ischaemic stroke (AIS) is caused by a severe blockage of an artery leading to immediate reduced blood flow to part of the brain. Standard therapies target the blocked artery by either dissolving the blockage or removing the blockage. However, even after successful treatment, re-blockage of arteries can occur. The use of an antiplatelet therapy, TBO-309, in addition to standard therapies offers the possibility of improved restoration of blood flow and reduced rates of artery re-blockage.

DETAILED DESCRIPTION:
Stroke is a leading cause of disability worldwide, with most strokes in Australia being Acute ischaemic stroke (AIS). AIS is caused by a severe blockage of an artery leading to immediate reduced blood flow to part of the brain. Timely restoration of blood flow is critical to preserve brain function. Standard therapies target the blocked artery by either dissolving the blockage (intravenous thrombolysis (IVT)) or removing the blockage (endovascular thrombectomy (EVT)). However, even after successful treatment, re-blockage of arteries can occur. The use of an antiplatelet therapy in addition to IVT/EVT offers the possibility of improved restoration of blood flow and reduced rates of artery re-blockage.

STARS is a prospective, multicentre, open-label, dose escalation, Phase IIa study to assess the safety and tolerability of TBO-309, an adjuvant antiplatelet therapy, in patients with AIS. The study will test the hypothesis that AIS patients who are treated with TBO-309 in conjunction with standard therapy (IVT alone or IVT + EVT) will not experience higher rates of ICH compared to the expected rates of ICH in patients treated with only standard therapy (IVT alone or IVT + EVT).

TBO-309 is a potent, selective and ATP competitive PI3Kβ inhibitor which blocks platelet activation adhesion/aggregation and promotes platelet disaggregation, thereby specifically inhibiting thrombosis without interfering with normal haemostasis. In order to evaluate safety at lower doses, four dose levels in total will be administered using a serial dose-escalation design. Doses will be assigned based on a dose escalation methodology commencing with lower doses assigned early in the study. As safety criteria are satisfied (based on ICH rates) doses will be increased. The dosage strength of TBO-309 to be administered (30mg, 60mg, 120mg or 180mg) will be assigned by the study database.

Patients presenting to hospital with an AIS will be assessed according to the trial inclusion and exclusion criteria by the Principal Investigator, or nominated delegate, on admission to the Emergency Department. Consent will be sought from either the patient or their Person Responsible/Medical Treatment Decision Maker prior to enrolment into the study. Standard therapy, either IVT alone or IVT + EVT, will commence and the TBO-309 will be administered at the same time as standard therapy. Following administration of study drug and treatment with standard therapies, patients will receive usual supportive care either in the Intensive Care Unit or in the hospital ward. Any significant neurological deterioration will require an emergency non-contrast CT head to assess for the presence of ICH. All patients will receive a 24-36 hour MRI or a multimodal CT to assess asymptomatic bleeding, recanalisation and infarct volume.

During the patients hospital stay clinical outcome data will be collected during the study period to document response to treatment and to monitor safety. Study patients will be followed-up for 90 days post-enrolment, or to death, whichever is the earlier.

ELIGIBILITY:
Inclusion Criteria

1. Patient aged 18 years or more
2. Patient has an acute ischaemic stroke
3. Patient will be treated with either:

   1. Intravenous thrombolysis (IVT) with alteplase or tenecteplase for a diagnosis of AIS that is confirmed by CT imaging;

      alone/OR WITH
   2. Endovascular Thrombectomy (EVT) for large vessel occlusion (LVO) in the internal carotid artery, middle cerebral artery (M1 segment), middle cerebral artery (M2 segment) or with tandem occlusion of both the cervical carotid and intracranial large arteries who either:

   i. presented within 6 hours of stroke onset

   OR

   ii. presented between 6-24 hours after they were last known to be well and clinical observations and either CT perfusion or MRI features indicate the presence of salvageable brain tissue, defined as ischaemic core <70mL with a mismatch ratio >1.8 and absolute mismatch >15mL.
4. Patient has at least a mild grade of neurological impairment i.e. NIHSS of 5 or more
5. Patient has an estimated pre-stroke mRS of less than 4

Exclusion Criteria

1. Patient is considered unlikely to benefit from study intervention defined by one of the following:

   1. Advanced dementia
   2. Severe pre-stroke disability (mRS score 4-5)
   3. Glasgow Coma Score (GCS) 3 to 5
   4. Evidence of a large well-defined ischaemic lesion measuring more than one third of the MCA territory
2. High likelihood of undergoing stent insertion and requiring additional antithrombotic(s)
3. Uncontrolled hypertension (SBP >180 or DBP >110, refractory to medical therapy)
4. ICH within the last 90 days
5. Myocardial infarction or stroke within the last 30 days
6. Patient has an underlying disease process with a life expectancy of <90 days
7. Contraindication to thrombolysis i.e. increased bleeding risk
8. Contraindication to intravenous contrast agents including renal impairment or allergy
9. Known treatment with dual antiplatelet therapy or anticoagulant medication
10. Known severe liver disease
11. Known bleeding disorder
12. Cardiopulmonary resuscitation or arterial puncture at non-compressible site or lumbar puncture within 7 days
13. Another medical illness or social circumstance that may interfere with outcome assessments and follow-up
14. Known or suspected pregnancy
15. Patients currently participating in another interventional clinical trial
16. Informed consent unable to be obtained from the patient or their Person Responsible/Medical Treatment Decision Maker prior to study interventions
17. Study drug cannot be given within one hour of thrombolytic drug bolus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with ICH within 24-36 hours of study drug (TBO-309) commencement. | Within 24-36 hours of initiation of study drug
  Proportion of patients with ICH within 24-36 hours of study drug (TBO-309) commencement. ICH is defined as parenchymal haemorrhage (PH) type II based on The Heidelberg Bleeding Classification or any intracranial haemorrhage leading to clinical deterioration i.e. an increase in NIHSS of 4 points or more, on post-intervention brain MRI with MRA or multimodal CT scan (see appendix 2 and 3). This definition allows the inclusion of any clinically and radiologically significant haemorrhage with the rate of expected ICH in this patient population estimated to be up to 8%

SECONDARY OUTCOMES:
All bleeding | Within 72 hours of study drug administration
  All bleeding within 72 hours of study drug (TBO-309) administration according to a modified WHO scale
All ICH | 24-36 hours
  All ICH demonstrated on 24-36 hours imaging (recommended in patients who did not have the 2-6 hours imaging)
All intracerebral hemorrhage (ICH) | Up to 90 days post study drug administration
  All ICH as demonstrated on CT/MRI up to 90 days
All bleeding | Up to 90 days post study drug administration
  All bleeding reported up to 90 days according to a modified WHO scale

OTHER OUTCOMES:
Recanalisation rate | Within 2-6 hours of study drug commencement
  CT Angiogram (CTA) or MR Angiogram (MRA) assessment 2-6 hours post study drug commencement in patients with visible vessel occlusion who do not receive endovascular thrombectomy to measure recanalisation rate by the Arterial Occlusive Lesion (AOL) scale
Reperfusion rates | Post EVT
  Reperfusion rates by expanded Thrombolysis in Cerebral Infarction scale (eTICI) 2b50 or better (i.e. 50% to 100%) at the initial catheter angiogram in patients receiving endovascular thrombectomy and at the end after patients have received endovascular thrombectomy.
Infarct volume | 24-36 hours post study drug commencement
  Infarct volume 24-36 hours post study drug commencement measured by Diffusion Weighted Imaging (DWI) MRI or CT scan
NIHSS score | At 24 hours, 72 hours and 7 days post study drug administration or hospital discharge (whichever is sooner)
  Quantifies stroke severity
Modified Rankin Scale (mRS) score | At hospital discharge and 90 days post study drug administration
  Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke.
Mortality | At 90 days post study drug administration
  All-cause mortality
Plasma levels of TBO-309 | At the end of infusion, and 1 and 3 hours post end of infusion
  Plasma levels of TBO-309 will be measured to generate a population pharmacokinetic model
AKT phosphorylation relative to total AKT | At the end of infusion
  AKT phosphorylation relative to total AKT (pAKT/AKT) from platelets at the end of infusion
Genomic markers | 24 hours post end of infusion
  Genomic markers of delayed TBO-309 clearance when individuals with delayed clearance are identified
Genetic markers for stroke outcome | 24 hours post end of infusion
  Putative genetic markers for stroke outcome, including bleeding and reperfusion, following TBO-309 administration

CONTACTS AND LOCATIONS:
Overall Officials: Candice Delcourt, Dr, Study Chair — The George Institute
Locations (7):
- Australia (7):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Eastern Health- Box Hill Hospital, Box Hill, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No